CLINICAL TRIAL: NCT00914407
Title: Measurement of Retinal Blood Flow, Retinal Oxygenation and Retinal Oxygen Extraction in Healthy Subjects During Normoxia and Systemic Hyperoxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. Priv.-Doz. Dr, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: OPHT-030209
Record Dates: First submitted 2009-06-04; First posted 2009-06-05 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Healthy; Normoxia; Systemic Hypoxia
Keywords: Ocular physiology
MeSH Terms: interventions — Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Healthy subjects (Experimental)
  Interventions: Drug: Oxygen

INTERVENTIONS:
Drug: Oxygen — 100% Oxygen inhalation for 30 minutes

SUMMARY:
The inner retina is crucially dependent on an adequate retinal blood supply. When the retina becomes ischemic and hypoxic this results in severe vision loss due to retinal neovascularization. Measurement of retinal blood flow and retinal oxygenation is, however, still a difficult task. Information on retinal oxygenation is almost unavailable from human studies. In the present protocol the investigators propose a procedure allowing for the measurement of retinal blood flow, retinal oxygenation and retinal oxygen extraction by combining a number of innovative techniques. Specifically, retinal vessel diameters will be measured with a Retinal Vessel Analyzer, retinal blood velocities with bi-directional laser Doppler velocimetry and retinal oxygenation with spectroscopic evaluation of retinal fundus images. This will allow for the calculation of retinal oxygen extraction, a fundamental parameter of retinal function. Up to now, no data for retinal oxygen extraction are available in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18 and 35 years
* Nonsmokers
* Body mass index between 15th and 85th percentile
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Normal laboratory values unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, ametropia < 3 Dpt

Exclusion Criteria:

* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Treatment in the previous 3 weeks with any drug except oral contraceptives
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Blood donation during the previous 3 weeks
* Pregnancy

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2010-04; Primary Completion 2016-12-10 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Retinal blood velocity Retinal vessel diameters Oxygen saturation of retinal vessels Oxygen extraction as calculated from these parameters | 20 min ocular blood flow measurement on 1 study day

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Fondi K, Aschinger GC, Bata AM, Wozniak PA, Liao L, Seidel G, Doblhoff-Dier V, Schmidl D, Garhofer G, Werkmeister RM, Schmetterer L. Measurement of Retinal Vascular Caliber From Optical Coherence Tomography Phase Images. Invest Ophthalmol Vis Sci. 2016 Jul 1;57(9):OCT121-9. doi: 10.1167/iovs.15-18476. PMID 27409462